CLINICAL TRIAL: NCT06023316
Title: mGain - sEMG-based Gamified Therapy for Improved Upper Limb Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: mGain-001
Record Dates: First submitted 2023-08-13; First posted 2023-09-05 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Upper Limb Weakness Due to Central Neurologic Injury; Upper Limb Weakness Due to Peripheral Neurologic Injury; Upper Limb Weakness Due to Nerve Reconstruction; Upper Limb Weakness Due to Tendon Transfer Surgery; Stroke; Upper Limb Amputation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- mGain system (Experimental): mGain system: passive, noninvasive, Bluetooth-enabled, wire-free, surface electromyography measurement device that provides input to a mobile app for an interactive gaming platform
  Interventions: Device: mGain system

INTERVENTIONS:
Device: mGain system — passive, noninvasive surface electromyography measurement device and gaming mobile application

SUMMARY:
The purpose of this Phase I study is to conduct a pilot clinical trial using a mobile app-connected, wire-free surface electromyography (sEMG) system, called mGain, that provides biofeedback-based therapy in individuals with upper limb weakness due to neurologic injury or with upper limb amputation. Our overarching hypothesis is that the mGain wireless sEMG device and mobile therapeutic gaming environment will demonstrate improved adherence to therapy when compared to standard of care and will be feasible, acceptable, and usable in individuals with upper limb weakness or limb amputation.

All participants will undertake four weeks of therapy. Conducting therapy five days a week for 30 minutes a day. In addition, participants will have an initial and final assessment visit at a study site, with each visit expected to last 1-2 hours.

DETAILED DESCRIPTION:
All participants will undertake four weeks of therapy. Conducting therapy five days a week for 30 minutes a day. In addition, participants will have an initial and final assessment visit at a study site, with each visit expected to last 1-2 hours.

Initial Assessment: Eligible individuals will complete a baseline assessment including range of motion, manual muscle testing, and handheld dynamometry of the target limb(s). Target muscles for therapy will be identified (e.g., biceps, triceps, deltoids, forearm flexors, forearm extensors) and a trial of sEMG evaluation to detect muscle signal will be conducted. If detectable muscle signal is present, participants will complete the consent process and be enrolled in the study. Each participant will be taught the use of the mGain system using their own mobile phone or tablet and be given a therapeutic regimen to target their individual muscle weakness. Participants will then be asked to demonstrate use of the system. Participants can ask questions to ensure they understand system usage and the expectations when at home. Participants will complete baseline validated outcome measures such as the QuickDASH (Disabilities of the Arm, Shoulder and Hand questionnaire) and PROMIS Self-Efficacy Scale.

Home Therapy: For the four weeks following the initial assessment, participants will be asked to conduct a minimum of 30 minutes of therapy per day, 5 days a week, at home using the mGain system targeting the muscles identified during the initial assessment. Individuals will be asked to complete short questionnaires and write in an eDiary about their experience after conducting their daily exercises. A member of the study team will contact the participants on a weekly basis to provide technical support, inquire about adherence, and encourage participation. Data for each participant will be uploaded to Orthocare Innovations' HIPAA compliant cloud-based server.

Final Assessment: Participants will complete a final assessment of strength, range of motion, and manual muscle testing. Additionally, participants will complete outcome measures and surveys such as the QuickDASH, PROMIS Self-Efficacy, system usability scale, and a custom feasibility survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Upper limb weakness due to central or peripheral neurologic injury, stroke, or nerve reconstruction or tendon transfer surgery within one year; or upper limb amputation (e.g., transradial or transhumeral)
* Muscle strength of three or less on the Medical Research Council Manual Muscle Testing grading scale in any of the following (as appropriate for individuals with intact limbs): shoulder abduction, elbow flexion, elbow extension, wrist extension, wrist flexion, or finger extension
* Access to and willingness to use smart phone or tablet
* Able to tolerate participation in activity for at least 30 minutes of therapy exercises per day for five days per week
* Able to provide written informed consent for study participation

Exclusion Criteria:

* Not able to read and understand English
* Pregnancy
* History of prior central or peripheral neurologic injury or neuromuscular condition
* No muscle activation detectable by the mGain sEMG sensor
* Progressive neurologic deficit
* Impaired dexterity on the contralateral side such that participant is unable to use the device
* Spasticity with modified Ashworth score of three or greater
* Severe joint contracture (>50% of available range)
* Sensitive skin that would not tolerate wearing the mGain sEMG sensor
* Medical instability
* Confounding injury, musculoskeletal issues, or cognitive issues that limit effective participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Pre Self-Efficacy | At initial assessment before using intervention
  The PROMIS Self-Efficacy is a validated patient-reported questionnaire that measures an individual's confidence in the ability to perform specific tasks or behaviors in a variety of situations; developed under the Patient-Reported Outcomes Measurement Information System (PROMIS) program; results in a T-score where 50 is the mean and T-scores below the mean indicate less self-efficacy.
Post Self-Efficacy | Four weeks (at final assessment after using intervention for four weeks)
  The PROMIS Self-Efficacy is a validated patient-reported questionnaire that measures an individual's confidence in the ability to perform specific tasks or behaviors in a variety of situations; developed under the Patient-Reported Outcomes Measurement Information System (PROMIS) program; results in a T-score where 50 is the mean and T-scores below the mean indicate less self-efficacy.
System Usability Scale | Four weeks (at final assessment after using intervention for four weeks)
  The System Usability Scale measures the usability of a system and is a 10-item questionnaire completed by the participant; results in score 0-100 where scores above 68 would be considered above average.

SECONDARY OUTCOMES:
pre-QuickDASH | At initial assessment before using intervention
  QuickDASH (Disabilities of the Arm, Shoulder and Hand) is a validated patient-reported questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb; results in score 0-100 where 0 represents the least disability and 100 represents the greatest disability
post-QuickDASH | Four weeks (at final assessment after using intervention for four weeks)
  QuickDASH is a validated patient-reported questionnaire that measures physical function and symptoms in people with musculoskeletal disorders of the upper limb; results in score 0-100 where 0 represents the least disability and 100 represents the greatest disability

CONTACTS AND LOCATIONS:
Overall Officials: David Boone, PhD, Principal Investigator — Orthocare Innovations, LLC
Locations (1):
- Orthocare Innovations, LLC, Edmonds, Washington, United States

IPD SHARING:
Plan to Share IPD: No